CLINICAL TRIAL: NCT03994991
Title: Personalized Neuromodulation for Treating Post-surgical Pain
Brief Title: Transcranial Magnetic Stimulation (TMS) for Thoracic Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We weren't able to enroll patients due to COVID19 pandemic.
Sponsor: Emine Bayman (Other)
Responsible Party: Sponsor-Investigator, Emine Bayman, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201906717
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Thoracic Surgery; Chronic Pain; Transcranial Magnetic Stimulation; Neuromodulation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be randomized to active TMS vs sham TMS groups with approximately a 2:1 ratio. At the end of the study, the investigators expect 24 patients to have active TMS and 12 patients to have sham TMS sessions.
  Patients in the sham TMS group will have appointments at the same time as the active TMS patients. The TMS device used for the sham TMS group patients will be identical to the active TMS group. Only the stimulation will be different.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TMS (Experimental): Patients in the active TMS group will receive active TMS 2 times a day for 5 days. In addition, these patients will have MRI before the first TMS session and after the last TMS session.
  Interventions: Device: active TMS
- Sham TMS (Sham Comparator): Patients in the shamTMS group will receive sham TMS 2 times a day for 5 days. In addition, these patients will have MRI before the first TMS session and after the last TMS session.
  Interventions: Device: sham TMS

INTERVENTIONS:
Device: active TMS — Transcranial magnetic stimulation
  Arms: Active TMS
Device: sham TMS — Sham transcranial magnetic stimulation
  Arms: Sham TMS

SUMMARY:
Patients with high severity of post-surgical pain scores will be randomized to transcranial magnetic stimulation (TMS) vs sham TMS groups. Both group of patients will have 10 TMS sessions during 5 days. Our hypothesis is that, the reduction in the severity of pain scores will be greater among those patients who are randomized to active TMS group compared to sham TMS group. The investigators will explore how improvements in pain correlate with changes in brain network connectivity.

DETAILED DESCRIPTION:
More than 25 million adults suffer from chronic pain in the United States making it the single most common symptom for which patients seek medical care. Although chronic pain can develop from a variety conditions, surgery is one of the most common and the incidence of chronic pain after thoracic surgery is particularly high. Opioids have been a mainstay therapy for post-surgical pain, but there is increasing awareness that post-surgical opioid use is a risk factor for addiction. Consequently, there are major nationwide efforts underway to limit opioid use in the post-surgical setting and identify safer options. One promising modality that has emerged in recent years is the use of non-invasive brain stimulation using transcranial magnetic stimulation (TMS).

TMS provides a method for noninvasively modulating cortical excitability, and a number of studies have shown that non-invasive neuromodulation can reduce pain in patients suffering from chronic pain. Using resting state functional magnetic resonance imaging, the investigators propose to investigate changes in brain networks after TMS and additionally investigate individual differences in brain network connectivity patterns that predict the effectiveness of TMS. The investigators expect that active TMS, compared to sham TMS, will normalize brain network connectivity and lead to lower pain and opioid use after surgery. In addition, by assessing pre-surgical brain networks, the investigators hope to identify brain connectivity patterns that predict efficacy of TMS as a post-surgical treatment option.

The investigators will recruit 36 subjects who've undergone thoracic surgery. The investigators will recruit primarily in-patients but may also recruit patients who have gone home after surgery.

During weeks 2-3 Post-Surgery, 5 study visits will be completed, each ranging in duration from 1 1/2 - 3 hours. All 5 visits include 2 short TMS sessions (10 total), pain and mood assessments. At V1 and V5, functional magnetic resonance imaging (fMRI) scans will be completed, as well as additional pain and health related assessments (many only done at V1). Also, short, follow-up phone calls will be completed at 3 and 6 months post-surgery to assess pain and other outcomes.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* 18 to 80 years old
* scheduled thoracic surgery w/one of the following procedures: thoracotomy, pneumonectomy, removal of lung other than bilobectomy, pneumonectomy, completion pneumonectomy, sleeve lobectomy, segmentectomy, single or multiple wedge resection, or thoracoscopy with excision-plication of bullae, with lobectomy, with partial or total pulmonary decortication or with wedge resection of lung.
* Post-surgery pain equal or greater 4 at phone screen

Exclusion Criteria:

* limitations of self-expression or visual dysfunction (as assessed by research team member during inpatient screen)
* having emergency surgery
* bipolar, schizophrenia or other psychotic disorders
* Alzheimer's, dementia, epilepsy, traumatic brain injury or other similarly impacting neurological issues
* pregnancy
* incarceration
* pain in thoracic region for last two or more months
* additional MRI/TMS exclusions: (implants, stents, neurostimulators, metal, claustrophobia, certain medications)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
The change in the severity of pain score after 5 days of active vs sham TMS. | 5 days
  The change in pain score will be calculated based on the following 2 pain scores:
  Day 1 NRS is the severity of pain collected at the beginning of the first study visit before the TMS and MRI sessions.
  Day 5 NRS is the severity of pain collected at the end of the 5th study visit, after the second TMS and the MRI session.
  The change in pain score is the difference between the day 5 NRS and the day 1 NRS.

SECONDARY OUTCOMES:
The presence of thoracic surgery related chronic pain at 6 months after surgery. | 6 months after thoracic surgery
  Pain assessments at 6 months aftger surgery will be made with phone interview. Patients will be asked if they still have pain related to their thoracic surgery ('Do you currently have pain related to your thoracic surgery? [yes/ no]')

CONTACTS AND LOCATIONS:
Overall Officials: Emine O Bayman, Principal Investigator — University of Iowa; Jatin Vaidya, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayman EO, Parekh KR, Keech J, Selte A, Brennan TJ. A Prospective Study of Chronic Pain after Thoracic Surgery. Anesthesiology. 2017 May;126(5):938-951. doi: 10.1097/ALN.0000000000001576. PMID 28248713
- [Background] Bayman EO, Parekh KR, Keech J, Larson N, Vander Weg M, Brennan TJ. Preoperative Patient Expectations of Postoperative Pain Are Associated with Moderate to Severe Acute Pain After VATS. Pain Med. 2019 Mar 1;20(3):543-554. doi: 10.1093/pm/pny096. PMID 29878248
- [Background] Bayman EO, Brennan TJ. Incidence and severity of chronic pain at 3 and 6 months after thoracotomy: meta-analysis. J Pain. 2014 Sep;15(9):887-97. doi: 10.1016/j.jpain.2014.06.005. Epub 2014 Jun 23. PMID 24968967